CLINICAL TRIAL: NCT06084234
Title: National Liver Cancer Screening Trial
Acronym: TRACER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other); University of Michigan (Other); Dana-Farber Cancer Institute (Other); Baylor College of Medicine (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Amit Singal, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TRACER; 2U24CA086368-22 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Hepatocellular; Liver Cancer; Liver Cirrhosis; Hepatitis B
Keywords: Hepatocellular carcinoma surveillance; GALAD; Alpha Fetoprotein
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Cirrhosis; Hepatitis B

STUDY DESIGN:
Intervention Model Description: This is a randomized open-label study comparing US ± AFP vs. GALAD-based surveillance every 6 (± 3-month window) months starting at randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A: Semi-annual surveillance using liver ultrasound +/- alpha-fetoprotein (Active Comparator): Participants in this arm will undergo current standard of care surveillance procedures i.e. liver ultrasound with or without alpha fetoprotein (AFP) measurement.
  Interventions: Diagnostic Test: Liver Ultrasound with or without AFP
- Arm B: Semi-annual surveillance using GALAD (Experimental): For participants in this arm, study team will order GALAD measurement every 6 months +/- 3 months.
  Interventions: Diagnostic Test: GALAD

INTERVENTIONS:
Diagnostic Test: GALAD — GALAD is a 3 biomarker panel incorporating AFP, AFP-L3% and DCP (all FDA approved), with patient age and sex.
  Arms: Arm B: Semi-annual surveillance using GALAD
Diagnostic Test: Liver Ultrasound with or without AFP — This intervention consists of current standard of care ultrasound based surveillance with or without alpha-fetoprotein measurement.
  Arms: Arm A: Semi-annual surveillance using liver ultrasound +/- alpha-fetoprotein

SUMMARY:
The National Liver Cancer Screening Trial is an adaptive randomized phase IV Trial comparing ultrasound-based versus biomarker-based screening in 5500 patients with cirrhosis from any etiology or patients with chronic hepatitis B infection. Eligible patients will be randomized in a 1:1 fashion to Arm A using semi-annual ultrasound and AFP-based screening or Arm B using semi-annual screening using GALAD alone. Randomization will be stratified by sex, enrolling site, Child Pugh class (A vs. B), and HCC etiology (viral vs. non-viral). Patients will be recruited from 15 sites (mix of tertiary care and large community health systems) over a 3-year period, and the primary endpoint of the phase IV trial, reduction in late-stage HCC, will be assessed after 5.5 years.

DETAILED DESCRIPTION:
The TRACER phase IV biomarker study is a randomized trial comparing ultrasound-based screening versus a biomarker-based strategy in patients with cirrhosis. In brief, 5500 patients with cirrhosis from any etiology would be randomized in a 1:1 fashion to Arm A offering semi-annual ultrasound +/- AFP-based screening or Arm B offering semi-annual biomarker-based screening. Randomization will be stratified by site, Child Pugh class (A vs. B), liver disease etiology (viral, non-viral, and non-cirrhotic HBV infection) and sex. Patients will be recruited from 15 sites (mix of tertiary care and large community health systems) over a 3-year period, and reduction in the proportion of late-stage HCC, will be assessed at the end of Year 5.5. If the results are promising, study team will continue extended follow-up and compare the incidence of late-stage HCC between the two arms at Year 8 and reduction in HCC mortality during long term follow up.

Study team will include adult patients, age ≥ 18 years, with Child Pugh class A or B cirrhosis of any etiology or non-cirrhotic chronic hepatitis B virus infection with PAGE-B score >9. Study team will exclude patients post liver transplantation, patients with Child Pugh C cirrhosis, patients with significant comorbidity and limited life expectancy, and those with history of other malignancy, except non-melanoma skin cancer or indolent tumors, within 3 years prior to enrollment given lack of screening recommendations in those patient populations. Study team will also exclude patients with suspicious liver masses at baseline as well as those with a solid lesion ≥1 cm on ultrasound or AFP ≥20 ng/mL without diagnostic evaluation to exclude HCC. Study team will also exclude patients in whom the provider plans to follow the patient with CT or MRI-based surveillance. GALAD is not recommended in patients with pregnancy or active warfarin use given known impact on biomarker performance, so these patients will be excluded.

At enrollment, study team will record patient demographics and clinical characteristics using a combination of electronic medical records and patient questionnaires. Patients will then be offered semi-annual surveillance as defined by their study arm: ultrasound and AFP for patients in Arm A and the biomarker, GALAD, for patients in Arm B. Repeat surveillance tests will be offered every six months (per assigned arm) for patients with normal surveillance results. Diagnostic evaluation with multi-phasic CT or contrast-enhanced MRI will be recommended for any patients with abnormal screening results. Patients with normal diagnostic testing (i.e., false positive result) will be recommended to return to their assigned surveillance arm. Standardized criteria from the AASLD and LI-RADS will be used to define incident HCC. Study team will use a set of validated surveys (e.g., Psychological Consequences Questionnaire, Decision Regret scale, FACIT-COST) to measure secondary outcomes of interest including psychological and financial harms.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet all of the following inclusion criteria:

1. Adult patients ages 18-85 with cirrhosis from any etiology or with chronic hepatitis B with a PAGE-B score greater than 9 within 12 months of enrollment
2. Patient is eligible for HCC surveillance according to treating physician or by the site investigator
3. Able to provide informed consent
4. Life expectancy >6 months (after consent) as determined by the treating provider or site investigator

Exclusion Criteria:

Patient will be excluded for any of the following exclusion criteria:

1. Child Pugh C cirrhosis
2. History or clinical symptoms of hepatocellular carcinoma or cholangiocarcinoma
3. History of solid nodule on baseline ultrasound (i.e., lesion 1cm or greater) within 9 months prior to consent without subsequent diagnostic CT/MRI demonstrating benign nature)
4. AFP >20 ng/mL within 6 months prior to consent, in the absence of a contrast-enhanced CT or MRI within 6 months of AFP (before or after) level demonstrating lack of suspicious liver lesions
5. Newly diagnosed LR-3 greater than or equal to 1 cm within 6 months prior to consent
6. History of LR-4, LR-5, or LR-M on multi-phase CT or contrast-enhanced MRI within 6 months prior to consent
7. Presence of another active cancer besides non-melanomatous skin cancer or indolent cancer under active surveillance (e.g., prostate cancer or renal cell carcinoma) within the 2 years prior to consent
8. Patient's provider is planning to use MRI- or CT- based surveillance moving forward
9. History of a transjugular intrahepatic portosystemic shunt (TIPS)
10. History of Fontan associated liver disease or cardiac cirrhosis
11. History of solid organ transplantation
12. Actively listed for liver transplantation
13. Diagnosis of alcohol-associated hepatitis within 3 months prior to consent
14. Documented current or continued signs and symptoms of acute Wilson disease (acute liver failure, acute neurological deficits, hemolysis)
15. In patients with primary sclerosing cholangitis (PSC): Current active cholangitis within 90 days prior to consent
16. Known or documented habitual non-adherence to previous research studies or medical procedures or unwillingness to adhere to protocol (e.g., unwilling to obtain consent or samples)
17. In patients living with HIV: CD4+ T cell count less than 100 cells/mm3 within 60 days prior to consent
18. Known pregnancy at consent
19. Active warfarin use

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5500 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HCC detected at late stage | 5.5 years
  Proportion of HCC detected at a late stage, defined as HCC beyond Milan Criteria (one tumor less than or equal to 5 cm or 2-3 tumors each less than or equal to 3 cm, in the absence of vascular invasion or extra-hepatic metastases)

SECONDARY OUTCOMES:
HCC Screening utilization | 5.5 years
  Defined as proportion time covered by screening; each completed screening test (US +/- AFP or GALAD) will provide up to six months of coverage (numerator) divided by the total follow-up for each patient.
Proportion of HCC detected at a late-stage (defined based on BCLC stage) | 5.5 years
  Defined as HCC beyond BCLC stage A (single tumor of any size without vascular invasion or extrahepatic spread; or 2-3 tumors equal to or less than 3 cm each, without vascular invasion or extrahepatic spread)
Incidence of late-stage HCC | 8 years
  Defined as incidence of HCC (extended follow-up) beyond Milan Criteria or BCLC stage A
Proportion of HCC cases that receive Curative therapy | 5.5 years
  Defined as count of participants in receipt of liver transplantation, surgical resection, local ablative therapy, or radiation segmentectomy
Number of participants who encountered screening related physical harm | 5.5 years
  Physical harms will be defined as count of participants in receipt of diagnostic imaging for false positive or indeterminate results.
Number of participants who encountered screening related financial harm | 5.5 years
  Financial harms will be defined by direct costs (charges for all screening and diagnostic testing and co-pays) and indirect costs (e.g., travel and lost wages)
Number of participants who encountered screening related Psychological harm | 5.5 years
  Count of participants who encountered Psychological harms that includes cancer-specific worry and decisional regret.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singal, MD, MS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (18):
- United States (18):
  - University of Southern California, Los Angeles, California
  - Stanford University, Redwood City, California
  - Kaiser Permanente, Roseville, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin Healthcare, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - The Feinstein Institutes, Northwell Health, Inc., Manhasset, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center and Parkland Hospital, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singal AG, Parikh ND, Kanwal F, Marrero JA, Deodhar S, Page-Lester S, Lopez C, Feng Z, Tayob N. National Liver Cancer Screening Trial (TRACER) study protocol. Hepatol Commun. 2024 Nov 4;8(11):e0565. doi: 10.1097/HC9.0000000000000565. eCollection 2024 Nov 1. PMID 39495136